CLINICAL TRIAL: NCT04040348
Title: A Phase I, Prospective, Open-label Trial to Evaluate the Safety, Tolerability and Exploratory Outcomes of Multiple Allogeneic Human Mesenchymal Stem Cells (HMSC) Infusions in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Alzheimer's Disease Stem Cells Multiple Infusions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bernard (Barry) Baumel (Other)
Responsible Party: Sponsor-Investigator, Bernard (Barry) Baumel, Assistant Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190438
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2023-07

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Stem cells; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- hMSC Treatment group (Experimental): Participants in the hMSC treatment group will receive a total of 4 doses of the hMSC intervention. Each dose will be administered once about every 13 weeks within a year period.
  Interventions: Biological: Approximately 100 million cells allogeneic hMSC

INTERVENTIONS:
Biological: Approximately 100 million cells allogeneic hMSC — Umbilical cord-derived, allogeneic hMSC administered intravenously at a dose of approximately 100 million cells per infusion.

SUMMARY:
The purpose of this research study is to test the safety, possible side effects, and possible effectiveness of mesenchymal stem cell infusions when given to people with a diagnosis of mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

All subjects enrolled in this trial must:

1. Provide written informed consent
2. Male or female subjects aged 50-85 years at time of signing Informed Consent
3. Mini-Mental State Examination (MMSE) between 20-26
4. Amyloid PET scan or CSF Aß1-42 positive for the presence of amyloid
5. Meet criteria for either Alzheimer's Disease or probable Alzheimer's Disease (AD) according to National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINDCDS/ARDRA)
6. Subjects, if taking cholinesterase inhibitor medications (donepezil, rivastigmine (oral or transdermal) or galantamine), are required to have been taking them on a stable dose for at least 3 months prior to Baseline Visit These medicines are not required
7. Subjects already taking memantine will not have an effect in the inclusion/exclusion criteria.
8. Have a study partner
9. No clinically significant abnormal screening laboratory values, as determined by the investigator
10. Women must be postmenopausal, surgically sterile, or having infertility. A postmenopausal woman is defined as either having an intact uterus with at least 12 months of spontaneous amenorrhea or a diagnosis of menopause, defined as an Follicular Stimulating Hormone (FSH) level of > 25 IU/L

Exclusion Criteria:

All subjects enrolled must not have:

1. Dementia other than AD
2. A negative Amyloid PET scan
3. Other neurodegenerative disease
4. Significant psychiatric illness (e.g., uncontrolled major depression, schizophrenia, bipolar affective disorder)
5. History of seizures
6. Contraindication for Magnetic Resonance Imaging (MRI)
7. History of malignancy, except:

   * > 5 years in remission prior to screening
   * Be excised or treated basal cell, squamous carcinoma or melanoma in situ
   * Prostate cancer in situ
   * Cervical carcinoma in situ
8. Uncontrolled medical conditions

   * Hypertension
   * Diabetes
   * Unstable angina or history of Myocardial Infarction (MI) within 1 year prior to screening
   * History of alcohol or drug use disorder (except tobacco use disorder) within 2 years before the screening visit
9. Brain MRI at screening that shows evidence of findings incompatible with a diagnosis of Alzheimer's disease. Volumetric MRI scans done within 6 months prior to ICF signature will be accepted if completed locally.
10. History of bleeding disorder
11. History of or positive results for Human Immunodeficiency Virus (HIV)
12. History of or positive results for Hepatitis C Virus (HCV) or Hepatitis B Virus (HBV)
13. Hypersensitivity to dimethyl sulfoxide (DMSO)
14. Inability to perform any of the assessments required for endpoint analysis
15. Currently receiving (or received within four weeks of screening) experimental agents for the treatment of AD or enrolled in clinical trials in the prior 3 months
16. Be a transplant recipient, or on active listing (or expected future listing) for transplant of any organ.
17. Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Number of Incidence of any Treatment-Emergent Serious Adverse Events (TE-SAEs) | One month post-infusion
  All adverse events will be evaluated by the investigator for relationship with the study intervention. Treatment-Emergent Serious Adverse Events is defined as any untoward medical occurrence with a reasonable possibility that it is caused by the study intervention that:
  * Is life-threatening (e.g.; leads to stroke or non-fatal pulmonary embolism);
  * Requires inpatient hospitalization or prolongation of existing hospitalization;
  * Results in persistent or significant disability/incapacity
  * Results in other clinically significant sign(s) or symptom(s), (e.g.; clinically asymptomatic brain microhemorrhages); or
  * Results in death

SECONDARY OUTCOMES:
Cognitive function over time as assessed by the Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog 11) | Up to Week 65
  The ADAS-Cog 11 is a 13-item version of ADAS-Cog comprising of the original 11-item ADAS-Cog as well as Delayed Recall and Digit Cancellation items. The total score ranges from 0-85 points, with a lower score indicating better performance.
Cognitive function over time as assessed by the Mini Mental State Examination (MMSE) of Folstein test | Up to Week 65
  The MMSE assesses orientation to time and place, immediate and delayed recall of words, attention and calculation, language (naming, comprehension and repetition), and spatial ability (copying a figure). The total score ranges from 0-30, with a higher score indicating better cognitive performance.
Depressive symptoms over time as assessed by the Geriatric Depression Scale (GDS) Short Version | Up to Week 65
  The GDS is a 15-item questionnaire with each item counting as one point. The total score ranges from 0 to 15 with a score greater than 5 indicating possible depression.
Participant quality of life over time assessed via Alzheimer's Disease Related Quality of Life (ADRQL-40) Questionnaire as completed by the caregiver | Up to Week 65
  ADRQL-40 is a questionnaire completed by the caregiver assessing the quality of life of the participant with AD. The total score for the ADRQL is computed by summing the values assigned to the responses, dividing the sum by the maximum value for the scale and multiplying the results by 100 to obtain a percentage score of 0 to 100. A higher score reflects a higher quality of life.
Participant quality of life over time as assessed via the Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Questionnaire as completed by the caregiver | Up to Week 65
  The ADCS-ADL is a 23 item questionnaire completed by the caregiver assessing the basic and instrumental activities of daily living by the AD participant. Total score range from 0-78 with the higher score indicating increased independence.
Neuropsychiatric Inventory-Q (NPI-Q) Scores over time | Up to Week 52
  The NPI-Q is a questionnaire used to assess behavioral changes common in dementia patients. This questionnaire is completed by the caregiver. The questionnaire consists of 12 items with each item having a scoring range between 0-3. The higher score indicates a more severe neuropsychiatric symptomatology.
Caregiver's Quality of life over time as assessed by the Caregiver Self-Assessment Questionnaire scores | Up to Week 52
  The Caregiver Self-Assessment questionnaire is completed by the caregiver. It is an 18-item questionnaire answered with a "yes" or "no". Evidence of distress is indicated for having over 10 "yes" answers.
Biomarker levels over time | Up to Week 65
  Serum blood inflammatory and biomarker levels will be evaluated including Interleukin-6 (IL-6), Neurofilament light (NfL), Amyloid Beta 40 (Aβ40) and Amyloid Beta 42 (Aβ42) in pg/mL.
Serum ApoE level over time | Up to Week 65
  Serum blood Apolipoprotein E (ApoE) will be evaluated in mg/dL.
Serum PRA level over time | Up to Week 65
  Serum blood Plasma Renin Activity (PRA) will be evaluated in ng/mL per hour.
Serum Tau protein level over time | Up to Week 65
  Serum blood Tau protein level will be evaluated in ng/L.
Cerebrospinal Fluid (CSF) Biomarker levels over time | Up to Week 52
  CSF inflammatory and biomarker levels will be evaluated including Interleukin-6 (IL-6), Neurofilament light (NfL), Amyloid Beta 40 (Aβ40) and Amyloid Beta 42 (Aβ42) in pg/mL.
CSF ApoE level over time | Up to Week 52
  CSF Apolipoprotein E (ApoE) levels will be evaluated in mg/dL.
CSF PRA level over time | Up to Week 52
  CSF Plasma Renin Activity (PRA) levels will be evaluated in ng/mL per hour.
CSF Tau protein level over time | Up to Week 52
  CSF Tau protein levels will be evaluated in ng/L.
Change in hippocampal volume | Baseline to Week 6, Baseline to Week 52
  Change in hippocampal volume will be assessed via MRI Brain volumetric studies

CONTACTS AND LOCATIONS:
Overall Officials: Bernard (Barry) Baumel, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No